CLINICAL TRIAL: NCT04210349
Title: Immunogenicity and Safety of the Shenzhen Quadrivalent Inactivated Influenza Vaccine Versus the Shenzhen Trivalent Inactivated Influenza Vaccine in Chinese Subjects From 6 Months of Age
Brief Title: Study of Shenzhen Quadrivalent Inactivated Influenza Vaccine Versus the Shenzhen Trivalent Inactivated Influenza Vaccine in Chinese Subjects From 6 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FSQ02; U1111-1174-4698 (Other: UTN)
Record Dates: First submitted 2019-11-26; First posted 2019-12-24 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Open-label (single arm for early safety review) in step 1. Modified double-blind in step 2 with an unblinded administrator used at each trial site. The administrator will not be involved in any of the blinded study assessments (e.g., safety).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group A: 6 to 35 months, previously unvaccinated, step 1 (Experimental): Participants will receive two injections of SP Shz QIV 0.5 mL at Day 0 and Day 28
  Interventions: Biological: Quadrivalent Influenza Vaccine
- Group 1: 6 to 35 months, step 2 (Experimental): Participants will receive one injection of SP Shz QIV 0.25 mL or SP Shz QIV 0.5 mL at Day 0 or SP Shz TIV1 0.25 mL or SP Shz TIV2 0.25 mL at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
  Interventions: Biological: Quadrivalent Influenza Vaccine; Biological: Trivalent Influenza Vaccine 1 SP Shz TIV1; Biological: Trivalent Influenza Vaccine 2 SP Shz TIV2
- Group 2: 3 to 8 years, step 2 (Experimental): Participants will receive one injection of SP Shz QIV 0.5 mL or SP Shz QIV 0.5 mL or SP Shz TIV1 0.5 mL or SP Shz TIV2 0.5 mL at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
  Interventions: Biological: Quadrivalent Influenza Vaccine; Biological: Trivalent Influenza Vaccine 1 SP Shz TIV1; Biological: Trivalent Influenza Vaccine 2 SP Shz TIV2
- Group 3: 9 to 17 years, step 2 (Experimental): Participants will receive one injection of SP Shz QIV 0.5 mL or SP Shz TIV1 0.5 mL or SP Shz TIV2 0.5 mL at Day 0.
  Interventions: Biological: Quadrivalent Influenza Vaccine; Biological: Trivalent Influenza Vaccine 1 SP Shz TIV1; Biological: Trivalent Influenza Vaccine 2 SP Shz TIV2
- Group 4: 18 to 60 years, step 2 (Experimental): Participants will receive one injection of SP Shz QIV 0.5 mL or SP Shz TIV1 0.5 mL or SP Shz TIV2 0.5 mL at Day 0.
  Interventions: Biological: Quadrivalent Influenza Vaccine; Biological: Trivalent Influenza Vaccine 1 SP Shz TIV1; Biological: Trivalent Influenza Vaccine 2 SP Shz TIV2
- Group 5: >=61 years (Experimental): Participants will receive one injection of SP Shz QIV 0.5 mL or SP Shz TIV1 0.5 mL or SP Shz TIV2 0.5 mL at Day 0.
  Interventions: Biological: Quadrivalent Influenza Vaccine; Biological: Trivalent Influenza Vaccine 1 SP Shz TIV1; Biological: Trivalent Influenza Vaccine 2 SP Shz TIV2

INTERVENTIONS:
Biological: Quadrivalent Influenza Vaccine — Pharmaceutical form: Suspension for injection Route of administration: intramuscular
Biological: Trivalent Influenza Vaccine 1 SP Shz TIV1 — Pharmaceutical form: Suspension for injection Route of administration: intramuscular
  Arms: Group 1: 6 to 35 months, step 2; Group 2: 3 to 8 years, step 2; Group 3: 9 to 17 years, step 2; Group 4: 18 to 60 years, step 2; Group 5: >=61 years
Biological: Trivalent Influenza Vaccine 2 SP Shz TIV2 — Pharmaceutical form: Suspension for injection Route of administration: intramuscular
  Arms: Group 1: 6 to 35 months, step 2; Group 2: 3 to 8 years, step 2; Group 3: 9 to 17 years, step 2; Group 4: 18 to 60 years, step 2; Group 5: >=61 years

SUMMARY:
The primary objectives of the study were:

* To demonstrate the non-inferiority of the immune response in terms of geometric mean titers (GMTs) and seroconversion rates of the SP Shz QIV compared with the SP Shz TIV containing the Victoria lineage strain (TIV1) and the SP Shz TIV containing the Yamagata lineage strain (TIV2) for each strain
* To describe the safety profile of each dosage of SP Shz QIV, TIV1 or TIV2

The secondary objectives of the study were:

* Group 1 (subjects 6-35 months): To demonstrate the superiority of the immune response of SP Shz QIV compared to TIV2 or TIV1 group after the last dose; demonstrate the superiority of the immune response of the 0.5 mL dose of SP Shz QIV compared to 0.25 mL dose of SP Shz QIV group after the last dose; describe the immune response after administration of the last dose of either SP Shz QIV or SP Shz TIV1 or SP Shz TIV2.
* Groups 2 through 5 (subjects ≥ 3 years): To demonstrate the superiority of the immune response of SP Shz QIV compared to TIV2 or TIV1 group after a single dose; describe the immune response after each and every dose for all subjects ≥ 3 years of either SP Shz QIV or SP Shz TIV1 or SP Shz TIV2
* Group 2 (subjects 3 to 8 years), previously unvaccinated ,receiving SP Shz QIV: To describe the immune response after administration of each dose of SP Shz QIV, first dose and second dose of SP Shz QIV respectively
* Group 5 (subjects ≥ 65 years only): To assess the compliance, in terms of immunogenicity, of SP Shz QIV with the requirements of the CHMP NfG CPMP/BWP/214/96 in subjects aged 65 years or older.
* To describe the safety profile of SP Shz QIV 0.5 mL after each dose.

DETAILED DESCRIPTION:
Study duration per participants approximately is 180 days

ELIGIBILITY:
Inclusion criteria :

* Aged ≥ 6 months on the day of the first study visit/inclusion
* In good health or with underlying medical condition(s) that are judged to be stable by the investigator. Medically-stable is defined as:

  * No new diagnosis OR
  * No new class of prescription drug initiated during the 3 months prior to enrollment
* For participants aged 6 months through 17 years: Informed consent form has been signed and dated by the parent(s) or another legally acceptable representative, if applicable. Additionally an assent form has been signed and dated by the subject if aged 8 through 17 years (based on local regulations). For subjects aged 18 years and above: Informed consent form has been signed and dated
* Subject / subject and parent/legally acceptable representative are able to attend all scheduled visits and to comply with all trial procedures
* For subjects aged 6 months to less than 12 months only: Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg

Exclusion criteria:

* Subject is pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination. To be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, or surgically sterile
* Participation at the time of study enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine or planned receipt of any vaccine within the period from 2 weeks before trial vaccination to 2 weeks following trial vaccination (or the last trial vaccination)
* For previously influenza vaccinated subjects: Previous vaccination against influenza (in the 2019-2020 season) with either the trial vaccine or another vaccine
* For previously influenza unvaccinated subjects: Any influenza vaccination (from birth to the day of inclusion) with either the trial vaccine or another vaccine
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Self-reported thrombocytopenia or known thrombocytopenia as reported by the parent/legally acceptable representative, contraindicating intramuscular (IM) vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Personal history of clinically significant developmental delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder
* Known seropositivity for human immunodeficiency virus, including known HIV carrier or patient
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (axillary temperature ≥ 37.1°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Personal history of Guillain-Barre syndrome
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7106 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titers of Influenza Antibodies for Subjects 6-35 months | 28 days post-final vaccination
  Geometric mean titers will be assessed by a hemagglutination (HAI) method
Participants Achieving Seroconversion Against Antigens for Subjects 6-35 months | 28 days post-final vaccination
  Influenza antibodies will be assessed using the HAI method.
Geometric Mean Titers of Antibodies for Subjects ≥ 3 years | Day 28
  Geometric mean titers will be assessed by a HAI method
Number of Participants Achieving Seroconversion Against Antigens for Subjects ≥ 3 years | Day 28
  Influenza antibodies will be assessed using the HAI method.
Number of Participants with Immediate Adverse Events | Within 30 minutes after vaccination
  Immediate adverse events includes unsolicited systemic adverse events occuring within 30 minutes after vaccination
Number of Participants With Solicited Injection Site or Systemic Reactions | Within 7 days after vaccination
  Injection site reactions: injection site tenderness/pain, erythema, swelling, induration, and ecchymosis. Systemic reactions: fever, vomiting, crying abnormal, drowsiness, appetite lost, and irritability for toddlers aged <= 23 months and fever, headache, malaise, myalgia and shivering for participants aged > 2 years.
Number of Participants with Unsolicited Adverse Events | Within 28 days after vaccination
  Adverse events other than solicited reactions
Number of Participants with Serious Adverse Events | From Day 0 to Day 56 for participants in Group A and from Day 0 to 6 months after last vaccination for participants in Group 1 through Group 5.
  Serious adverse events (including adverse event of special interest) are assessed throughout the study.

SECONDARY OUTCOMES:
Geometric Mean Titers of Antibodies | Day 0 and 28 days post-final vaccination
  Geometric mean titers will be assessed by a HAI method.
Geometric Mean Individual Titer Ratio | Day 0 and 28 days post-final vaccination
  Geometric mean titers will be assessed by a HAI method.
Number of Participants with Detectable Titer ≥ 10 (1/dilution [1/dil]) | Day 0 and 28 days post-final vaccination
  Geometric mean titers will be assessed by an HAI method.
Percentage of Participants with Seroprotection to Antigens After Vaccination | Day 0 and 28 days post-final vaccination
  Seroprotection was defined as antibody titer ≥ 40 (1/dil) on Day 0 and on 28 days post-final vaccination
Percentage of Participants with Seroconversion to Antigens After Vaccination | Day 0 and 28 days post-final vaccination
  Seroconversion titer < 10 (1/dil) on Day 0 and post-injection(s) titer ≥ 40 (1/dil) on Day 28 or Day 56, or titer ≥ 10 (1/dil) on Day 0 and ≥ 4-fold increase of post-injection(s) titer on 28 days post-final vaccination.
Geometric Mean Individual Titer Ratio for Participants Aged 65 years or Older | Day 0 and 28 days post-final vaccination
  Geometric mean titers will be assessed by an HAI method.
Percentage of Participants with Seroconversion to Antigens After Vaccination for Participants Aged 65 years or Older | Day 0 and 28 days post-final vaccination
  Seroconversion titer < 10 (1/dil) on Day 0 and post-injection(s) titer ≥ 40 (1/dil) on Day 28, or titer ≥ 10 (1/dil) on Day 0 and ≥ 4-fold increase of post-injection(s) titer on 28 days post-final vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (7):
- China (7):
  - Investigational Site Number 1561000, Kunming
  - Investigational Site Number 1561001, Lincang
  - Investigational Site Number 1561002, Lincang
  - Investigational Site Number 1561003, Lincang
  - Investigational Site Number 1562001, Shangqiu
  - Investigational Site Number 1562002, Xinxiang
  - Investigational Site Number 1562000, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Liu X, Park J, Xia S, Liang B, Yang S, Wang Y, Syrkina O, Lavis N, Liu S, Zhao C, Ding J, Hu J, Samson SI, de Bruijn IA; FSQ01 and FSQ02 Study Groups. Immunological non-inferiority and safety of a quadrivalent inactivated influenza vaccine versus two trivalent inactivated influenza vaccines in China: Results from two studies. Hum Vaccin Immunother. 2022 Nov 30;18(6):2132798. doi: 10.1080/21645515.2022.2132798. Epub 2022 Nov 3. PMID 36328438
- See also: FSQ02 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25268&tenant=MT_SNY_9011